CLINICAL TRIAL: NCT06691295
Title: Exploring Transdiagnostic Psychological Processes in Functional Neurological Disorder
Acronym: Process-TNF
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 23-5173
Record Dates: First submitted 2024-11-12; First posted 2024-11-15 (Actual); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Functionnal Neurological Disorder
Keywords: Functional neurological disorder Transdiagnostic psychological processes
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with functional neurological disorders.: This study focuses on adult subjects with newly diagnosed functional neurological disorders (less than 5 years old) and prior to therapeutic management.
  Interventions: Other: Questionnaires

INTERVENTIONS:
Other: Questionnaires — This study aims to explore transdiagnostic psychological processes (PP) via the administration of self-reported scales and questionnaires, in a population of newly diagnosed FND patients, prior to any therapeutic management.
  The main objective is to describe the psychometric properties (scores on tools measuring psychological processes) of NFT patients (presenting the main phenotypes; sensitivo-motor; and seizures and discomfort).

SUMMARY:
Functional neurological disorder (FND) is a little-known borderline disorder between psychiatry and neurology, which is benefiting from renewed research. Characterized by neurological symptoms in the absence of lesion damage corresponding to the symptom, the disorder is thought to be due to functional impairment of the central nervous system (DSM5 American Psychiatric Association, 2013). Symptoms are non-congruent, discordant and inconsistent with current anatomical knowledge. Several phenotypes are listed and may be associated: among the most frequent are motor and sensory disorders and dissociative crises or seizures.

Common (Carson & Lehn, 2016) and disabling (Gendre et al., 2019), the neurobiological and psychological mechanisms involved in NFT are becoming better understood, yet its etiology remains enigmatic (Hallett et al., 2022). Recent theoretical models consider neuropsychological constructs as central to the development and maintenance of the disorder, influenced by emotional processes (Drane et al., 2020).

With a reputation for being difficult to treat, FND is a clinical challenge, and cognitive-behavioural therapy (CBT), although advocated, shows limits of efficacy mainly due to the complexity of clinical pictures and the heterogeneity of profiles (Gutkin et al., 2021). The CBTs described for FND are not specific to the disorder, and do not appear to be developed around a general theoretical framework defining the psychological mechanisms of the disorder (Richardson et al., 2020).

Thus, there would be an interest in identifying characteristics in these patients that could guide therapeutic choices and implement a better therapeutic response (Gutkin et al., 2021). These findings, coupled with the growing interest in this complex disorder, confirm the need to deepen our knowledge of the psychological mechanisms involved in the disorder, with a view to developing and testing a specialized and flexible clinic (Aybek et al., 2020).

Given the complexity of the disorder, a transdiagnostic approach is suggested (Saxena & Perez, 2021). The transdiagnostic processual approach (Harvey et al., 2004) proposes an innovative conceptualization of mental health problems. This model sees the human biological system as leading to psychological disorder through the disruption of initially normal psychological processes (Kinderman, 2005). These processes refer to psychological mechanisms on which the clinician can act, via validated therapeutic strategies. Transdiagnostic treatments apply the same underlying treatment principles to all mental disorders, without tailoring the protocol to specific diagnoses (Menon et al., 2017).

Considering the psychological mechanisms described as being altered in the disorder, etiological hypotheses, and literature data concerning transdiagnostic psychological processes, we raise the question of the involvement of such processes in FND. The aim of this study is to explore these processes in an FND population, with a view to refining our understanding of the psychological profile of these patients and guiding treatment.

ELIGIBILITY:
* Inclusion Criteria * :

  * Subjects diagnosed with FND by a neurologist ("Conversion disorder (disorder with functional neurological symptomatology" in DSM5)) from neurological report
  * Subject presenting one of the main phenotypes, i.e. 1. sensitivo-motor, 2. seizure / malaise (CNEP) as indicated by neurological report
  * Prior to any psychological, psychiatric or rehabilitative treatment for this TNF
  * Subject able to receive information and not to object to the use of his/her data for research purposes
* Exclusion Criteria * :

  * Subjects with symptoms corresponding to a pure pain or cognitive phenotype - patient's medical record
  * Subject with cognitive disorders - Moca score < 18
  * Subjects with diagnosed psychiatric comorbidities according to psychiatric CR + HADS scores A > 11 and D > 11
  * Subjects with neurological comorbidities - according to neurologist's CR

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort is selected from patients in the PULS-TNF program, which takes in all FND patients from the university hospital of Lyon or referred by other physicians.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-07-07 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Uncertainty Intolerance Scale - II | Data collected from May to July 2024 at the time of patient integration into the specialized FND care pathway.
  Scores on the Uncertainty Intolerance Scale - II to assess intolerance of uncertainty.
Metacognitive Belief Questionnaire - MCQ-30 | Data collected from May to July 2024 at the time of patient integration into the specialized FND care pathway.
  Scores on the Metacognitive Belief Questionnaire - MCQ-30 to assess metacognitive beliefs.
Ruminations Scale - Mini-CERTS | Data collected from May to July 2024 at the time of patient integration into the specialized FND care pathway.
  Scores on the Ruminations Scale - Mini-CERTS to assess ruminative thinking patterns.
Experiential Avoidance Questionnaire - MEAQ-short | Data collected from May to July 2024 at the time of patient integration into the specialized FND care pathway.
  Scores on the Experiential Avoidance Questionnaire - MEAQ-short to assess experiential avoidance.
Personalized Psychological Flexibility Index - PPFI | Data collected from May to July 2024 at the time of patient integration into the specialized FND care pathway.
  Scores on the Personalized Psychological Flexibility Index - PPFI to assess psychological flexibility.
Emotional Regulation Scale - DERS-F | Data collected from May to July 2024 at the time of patient integration into the specialized FND care pathway.
  Scores on the Emotional Regulation Scale - DERS-F to assess emotional regulation.
Somatoform Dissociation Questionnaire - SDQ-20 | Data collected from May to July 2024 at the time of patient integration into the specialized FND care pathway.
  Scores on the Somatoform Dissociation Questionnaire - SDQ-20 to assess somatoform dissociation.
Short Form Health Survey - SF-36 | Data collected from May to July 2024 at the time of patient integration into the specialized FND care pathway.
  Scores on the Short Form Health Survey - SF-36 to assess general health and quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: BOUAMMARI Annablle, Principal Investigator — Neurologie inflammatoire Hôpital P. Wertheimer/GHE
Locations (1):
- Hopital Pierre Wertheimer, Bron, France